CLINICAL TRIAL: NCT04204434
Title: Biomarkers For Immune Checkpoint Inhibitors
Status: Completed | Type: Observational
Sponsor: Rhode Island Hospital (Other)
Collaborators: Brown University (Other)
Responsible Party: Sponsor
Other Study IDs: Biomarkers For I.C. Inhibitors
Record Dates: First submitted 2016-08-16; First posted 2019-12-19 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-02

CONDITIONS: Advanced Cancer; Neoplasms
Keywords: Cancer; Advanced; Solid Tumor; Advanced Solid Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Stool, tissue, blood, and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a laboratory, non-treatment study. Immune checkpoint inhibitors are a type of immunotherapy that stimulates a patients immune system to fight their cancer. Immune checkpoint inhibitors are standard, FDA approved treatment for certain types of cancers such as melanoma, lung cancer, kidney cancer and bladder cancer. The laboratories of Dr. Jack Elias and Dr. Chun Geun Lee at Brown University are studying how immune checkpoint inhibitors work.Kintai Therapeutics is a biotech company in Cambridge Massachusetts that will focus on the molecules present in the GI tract, including the stomach, small intestine and colon.

DETAILED DESCRIPTION:
Patients who are receiving immune checkpoint inhibitors for their cancer treatment are eligible. Patients will sign informed consent. Ten cc of blood will be drawn before beginning immune checkpoint inhibitors and 10 cc of blood will be drawn 1-4 months after treatment is initiated. Deidentitified blood samples will be sent to the lab of Dr. Jack Elias and Dr. Chun Geul Lee and analyzed for biomarkers. The blood samples will be linked to the patient by a research number. Response to treatment will be correlated to potential biomarkers. The stool samples will be linked to the patient by a research number. Bacterial DNA and RNA may be sequenced and data used to identify bacterial taxa and genes within the stool. In compliance with NIH guidelines, all human DNA data would be removed computationally, and will not be used in any analyses. Small molecules may be profiled with metabolomics. Bacteria may also be isolated from the stool into in vitro culture, and efficacy of single-strains or communities and/or their DNA, RNA, and metabolites on disease models may be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced solid tumors initiating treatment with an immune checkpoint inhibitor.
* No prior immune checkpoint inhibitors
* Age >18.
* Signed informed consent

Exclusion Criteria:

* The patient is unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with an advanced solid cancer prior to initiating treatment with an immune checkpoint inhibitor are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
To determine serum predictors of response to immune checkpoint inhibitors at study entry, prior to checkpoint inhibitor therapy | At study entry, prior to checkpoint inhibitor therapy Anytime between 6-12 weeks after initiating treatment.
  Measure biomarker levels of immune checkpoint inhibitors in blood serum
To determine serum predictors of response to immune checkpoint inhibitors 4-weeks after initiation of treatment | Within 4 weeks after initiation of treatment
  Measure biomarker levels of immune checkpoint inhibitorsin blood serum
To determine serum predictors of response to immune checkpoint inhibitors anytime between 6-12 weeks after initiating treatment. | 6-12 weeks after initiating treatment
  Measure biomarker levels of immune checkpoint inhibitors in blood serum

SECONDARY OUTCOMES:
To evaluate bacteria, and bacterial products in gut microbiome before and after treatment with immune checkpoint inhibitors and correlate to response and toxicity. | At study entry, prior to immune checkpoint inhibitor therapy
  Measure bacteria and bacterial products in gut micobiome
To evaluate bacteria, and bacterial products in gut microbiome before and after treatment with immune checkpoint inhibitors and correlate to response and toxicity. | Within 4 weeks after initiation of treatment
  Measure bacteria and bacterial products in gut micobiome
To evaluate bacteria, and bacterial products in gut microbiome before and after treatment with immune checkpoint inhibitors and correlate to response and toxicity. | Anytime between 6-12 weeks after initiating treatment.
  Measure bacteria and bacterial products in gut micobiome

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — Rhode Island Hospital
Locations (2):
- United States (2):
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fife BT, Pauken KE. The role of the PD-1 pathway in autoimmunity and peripheral tolerance. Ann N Y Acad Sci. 2011 Jan;1217:45-59. doi: 10.1111/j.1749-6632.2010.05919.x. PMID 21276005
- [Background] Riley JL. PD-1 signaling in primary T cells. Immunol Rev. 2009 May;229(1):114-25. doi: 10.1111/j.1600-065X.2009.00767.x. PMID 19426218
- [Background] Doi T, Piha-Paul SA, Jalal SI, et al. Pembrolizumab (MK-3475) for patients with advanced esophageal carcinoma: Preliminary results from KEYNOTE-028.J Clin Oncol 33, 2015 (suppl; abstr 4010).
- [Background] Hamid O, Robert C, Daud A, Hodi FS, Hwu WJ, Kefford R, Wolchok JD, Hersey P, Joseph RW, Weber JS, Dronca R, Gangadhar TC, Patnaik A, Zarour H, Joshua AM, Gergich K, Elassaiss-Schaap J, Algazi A, Mateus C, Boasberg P, Tumeh PC, Chmielowski B, Ebbinghaus SW, Li XN, Kang SP, Ribas A. Safety and tumor responses with lambrolizumab (anti-PD-1) in melanoma. N Engl J Med. 2013 Jul 11;369(2):134-44. doi: 10.1056/NEJMoa1305133. Epub 2013 Jun 2. PMID 23724846
- [Background] Le D, Bendell JC, Calvo E, et al. Safety and activity of nivolumab monotherapy in advanced and metastatic (A/M) gastric or gastroesophageal junction cancer (GC/GEC): Results from the CheckMate-032 study. J Clin Oncol 34; 2016 (supp; abstr 06).
- [Background] Motzer RJ, Rini BI, McDermott DF, Redman BG, Kuzel TM, Harrison MR, Vaishampayan UN, Drabkin HA, George S, Logan TF, Margolin KA, Plimack ER, Lambert AM, Waxman IM, Hammers HJ. Nivolumab for Metastatic Renal Cell Carcinoma: Results of a Randomized Phase II Trial. J Clin Oncol. 2015 May 1;33(13):1430-7. doi: 10.1200/JCO.2014.59.0703. Epub 2014 Dec 1. PMID 25452452
- [Background] Patnaik A, Kang SP, Rasco D, Papadopoulos KP, Elassaiss-Schaap J, Beeram M, Drengler R, Chen C, Smith L, Espino G, Gergich K, Delgado L, Daud A, Lindia JA, Li XN, Pierce RH, Yearley JH, Wu D, Laterza O, Lehnert M, Iannone R, Tolcher AW. Phase I Study of Pembrolizumab (MK-3475; Anti-PD-1 Monoclonal Antibody) in Patients with Advanced Solid Tumors. Clin Cancer Res. 2015 Oct 1;21(19):4286-93. doi: 10.1158/1078-0432.CCR-14-2607. Epub 2015 May 14. PMID 25977344
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Durham NM, Nirschl CJ, Jackson CM, Elias J, Kochel CM, Anders RA, Drake CG. Lymphocyte Activation Gene 3 (LAG-3) modulates the ability of CD4 T-cells to be suppressed in vivo. PLoS One. 2014 Nov 5;9(11):e109080. doi: 10.1371/journal.pone.0109080. eCollection 2014. PMID 25372844
- [Background] Lee CM, He CH, Nour AM, Zhou Y, Ma B, Park JW, Kim KH, Dela Cruz C, Sharma L, Nasr ML, Modis Y, Lee CG, Elias JA. IL-13Ralpha2 uses TMEM219 in chitinase 3-like-1-induced signalling and effector responses. Nat Commun. 2016 Sep 15;7:12752. doi: 10.1038/ncomms12752. PMID 27629921
- [Background] Routy B, Le Chatelier E, Derosa L, Duong CPM, Alou MT, Daillere R, Fluckiger A, Messaoudene M, Rauber C, Roberti MP, Fidelle M, Flament C, Poirier-Colame V, Opolon P, Klein C, Iribarren K, Mondragon L, Jacquelot N, Qu B, Ferrere G, Clemenson C, Mezquita L, Masip JR, Naltet C, Brosseau S, Kaderbhai C, Richard C, Rizvi H, Levenez F, Galleron N, Quinquis B, Pons N, Ryffel B, Minard-Colin V, Gonin P, Soria JC, Deutsch E, Loriot Y, Ghiringhelli F, Zalcman G, Goldwasser F, Escudier B, Hellmann MD, Eggermont A, Raoult D, Albiges L, Kroemer G, Zitvogel L. Gut microbiome influences efficacy of PD-1-based immunotherapy against epithelial tumors. Science. 2018 Jan 5;359(6371):91-97. doi: 10.1126/science.aan3706. Epub 2017 Nov 2. PMID 29097494
- [Background] Pernot S, Ramtohul T, Taieb J. Checkpoint inhibitors and gastrointestinal immune-related adverse events. Curr Opin Oncol. 2016 Jul;28(4):264-8. doi: 10.1097/CCO.0000000000000292. PMID 27138569
- [Result] Latchman Y, Wood CR, Chernova T, Chaudhary D, Borde M, Chernova I, Iwai Y, Long AJ, Brown JA, Nunes R, Greenfield EA, Bourque K, Boussiotis VA, Carter LL, Carreno BM, Malenkovich N, Nishimura H, Okazaki T, Honjo T, Sharpe AH, Freeman GJ. PD-L2 is a second ligand for PD-1 and inhibits T cell activation. Nat Immunol. 2001 Mar;2(3):261-8. doi: 10.1038/85330. PMID 11224527